CLINICAL TRIAL: NCT07135908
Title: Assistant Professor
Brief Title: The Effect of the Solution-Focused Approach on Social Participation Skills and Hope in Children Living in Residential Care Objective: This Study Aimed to Evaluate the Effect of a Solution-focused Approach Program on the Hope Levels and Social Participation Skills of Children Living in Institutional
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Fatih Sahin, Assistant Professor, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 128676
Record Dates: First submitted 2025-07-27; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Hope; Nursing; Social Acceptance
Keywords: hope; Mental Health Care; Child Welfare; Psychosocial intervention; Nursing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Solution-Focused Approach Program) (Experimental): After the data collection tools were administered to the students, the Solution-Focused Approach Program was implemented with the experimental group students by the researcher for six weeks, one day per week for 60 minutes per day. The content of the Solution-Focused Approach Program was prepared in accordance with literature and reviewed by experts. The program content is as follows.
  Week: Introduction and informing the group
  Week: Understanding the importance of communication, being able to use active listening skills as an element of communication skills, establishing empathetic communication
  Week: Understanding the importance of social participation and identifying realistic hopes for the future
  Week: Becoming aware of sources of social participation and hope, creating mental maps for coping techniques and solutions
  Week: Drawing attention to change, gaining awareness, focusing on solutions, acquiring problem-solving skills
  Week: Ending the process, evaluating the process,
  Interventions: Behavioral: solution-oriented approach
- control group (No Intervention (Usual Care at Residential Institution) (No Intervention): No specific intervention was implemented in this group.

INTERVENTIONS:
Behavioral: solution-oriented approach — In this study, the solution-focused intervention was a structured psychosocial support program based on the principles of Solution-Focused Brief Therapy (SFBT). It consisted of six weekly sessions, each lasting 60 minutes, and was designed to help institutionalized children improve their hope levels and social participation skills.
  The sessions included:
  Enhancing communication and interpersonal skills
  Identifying personal strengths and sources of hope
  Developing social engagement strategies
  Teaching simple problem-solving techniques
  The approach focused on children's existing resources and future goals rather than their past problems. It encouraged positive thinking, goal setting, and active participation, promoting emotional resilience and social functioning.
  Arms: experimental group (Solution-Focused Approach Program)

SUMMARY:
his study examined whether a solution-focused approach program could improve hope and social participation skills in children living in institutional care. A total of 57 children were included and randomly divided into intervention and control groups. The intervention group attended a 6-week program with weekly 60-minute sessions focusing on communication, social skills, hope-building, and problem-solving.

The aim was to explore the potential applicability of solution-focused interventions in supporting the psychosocial development of institutionalized children within psychiatric nursing and caregiving practices.

DETAILED DESCRIPTION:
What Was the Purpose of This Study? To evaluate whether a solution-focused approach program could improve hope levels and social participation skills in children living in institutional care.

Who Participated? A total of 57 children living in a government care institution took part in the study. They were randomly assigned to intervention and control groups.

What Was Done?

The intervention group received a 6-week program based on solution-focused therapy. Each session lasted 60 minutes and included:

Communication skills

Social participation

Identifying sources of hope

Problem-solving techniques

What Were the Results? The study aimed to assess potential changes in hope and social skills among children participating in the program compared to those who did not.

Why Is This Important? Solution-focused methods may offer a structured framework for supporting the mental health and social development of children in institutional care. Such approaches could be adapted by nurses, social workers, and care staff in similar settings.

ELIGIBILITY:
Inclusion Criteria:

* To be residing in child care homes,
* To be continuing their education,
* To have no problems with hearing or visual abilities.

Exclusion Criteria:

those who did not meet the inclusion criteria

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
pretest (6-week solution-focused approach before the intervention) | Baseline (1 week before intervention)
  Primary Outcome Measure 1: Hope Level at Baseline (Children's Hope Scale)
  Description: The Children's Hope Scale (CHS) is a 6-item self-report tool assessing children's hopeful thinking. Scores range from 6 to 36; higher scores indicate greater hope.
  Time Frame: Baseline (within 1 week before intervention).
  Unit of Measure: Total score (6-36).
pretest pretest (6-week solution-focused approach before the intervention) | Baseline (within 1 week before intervention).
  Primary Outcome Measure 2: Social Participation Skills at Baseline (Social Skills Scale)
  Description: The Social Skills Rating System - Social Skills Scale (SSRS) evaluates cooperation, assertion, empathy, and self-control. Scores range from 0 to 90; higher scores indicate better functioning.
  Time Frame: Baseline (within 1 week before intervention).
  Unit of Measure: Total score (0-90).

SECONDARY OUTCOMES:
posttest (After the 6-week solution-focused approach intervention) | 6 weeks after baseline (post-intervention)
  Secondary Outcome Measure 1: Hope Level at Post-Test (Children's Hope Scale)
  Description: The Children's Hope Scale (CHS) is a 6-item self-report tool assessing children's hopeful thinking. Scores range from 6 to 36; higher scores indicate greater hope.
  Time Frame: Post-intervention (6 weeks after completion of the intervention).
  Unit of Measure: Total score (6-36).
posttest (After the 6-week solution-focused approach intervention) | Time Frame: Post-intervention (6 weeks after completion of the intervention).
  Secondary Outcome Measure 2: Social Participation Skills at Post-Test (Social Skills Scale)
  Description: The Social Skills Rating System - Social Skills Scale (SSRS) evaluates cooperation, assertion, empathy, and self-control. Scores range from 0 to 90; higher scores indicate better functioning.
  Time Frame: Post-intervention (6 weeks after completion of the intervention).
  Unit of Measure: Total score (0-90).

CONTACTS AND LOCATIONS:
Overall Officials: fatih şahin, dr, Principal Investigator — https://www.alparslan.edu.tr/tr
Locations (1):
- Aile Ve Sosyal Hizmetler Il Müdürlüğü, Muş, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.aile.gov.tr/mus